CLINICAL TRIAL: NCT07276061
Title: Outpatient Total Knee Prosthesis, Comparison of Postoperative Recovery Versus Conventional Hospitalization: a Retrospective, Single-center, Observational, Comparative Study of Superiority
Brief Title: Outpatient Total Knee Arthroscopy (TKA): Comparison of Postoperative Recovery Versus a Conventional Hospitalization
Acronym: PTG
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9240
Record Dates: First submitted 2025-03-25; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Knee Arthroscopy
Keywords: knee arthroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Outpatient TKA is a controversial topic due to concerns about its safety as an outpatient procedure, and remains a marginal procedure. Advances in enhanced postoperative rehabilitation protocols, coupled with advances in minimally invasive surgery, have made it possible to operate on an increasing number of patients on an outpatient basis. However, there are no studies in the literature analyzing functional recovery after outpatient TKA in France. The objective of this study was to compare postoperative recovery, assessed by the QoR-15F score, in patients undergoing outpatient TKA compared to those undergoing a conventional hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older (no upper age limit)
* Undergoing scheduled unilateral total knee replacement surgery between January 1, 2020 and June 30, 2023 at the Strasbourg University Hospitals
* Assessed using the QoR-15F score

Exclusion Criteria:

* Subject who has expressed opposition to the reuse of their data for scientific research purposes.
* Revision, emergency, oncological, bilateral, or septic surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female, 18 years of age or older (no upper age limit) undergoing scheduled unilateral total knee replacement surgery between January 1, 2020 and June 30, 2023 at the Strasbourg University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
QoR-15F score | at Day 1,Day 3, Day 14 and Day 28 post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie - Réanimation & Médecine Périopératoire - CHU de Strasbourg - France, Strasbourg, France